CLINICAL TRIAL: NCT01017393
Title: Preemptive Low-dose Epidural Ketamine for Preventing Chronic Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JHBahk_epidural ketamine PTPS
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Post-thoracotomy Pain
Keywords: preemptive epidural ketamine; prevention of chronic post-thoracotomy pain
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- ketamine (Experimental): epidural ketamine added to the patient controlled epidural analgesia regimen
  Interventions: Drug: Ketamine
- ketamine free (Active Comparator): epidural ketamine NOT added to the patient controlled epidural analgesia regimen
  Interventions: Drug: ketamine free

INTERVENTIONS:
Drug: Ketamine
  Arms: ketamine
Drug: ketamine free
  Arms: ketamine free

SUMMARY:
Chronic post-thoracotomy pain is the most common long-term complication that occurs after a thoracotomy with a reported incidence of up to 80%. While thoracic epidural analgesia has become the mainstay for managing acute post-thoracotomy pain, its effect on the chronic post-thoracotomy pain seems questionable. The objective of this prospective, double-blinded, randomized, controlled trial was to assess the effect of preemptive low-dose epidural ketamine in addition to preemptive thoracic epidural analgesia on the incidence of chronic post-thoracotomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery with a thoracotomy incision

Exclusion Criteria:

* history of previous thoracic surgery, chronic pain, psychiatric disease, cardiac or vascular disease, neurologic deficits, or contraindications to epidural catheterization such as coagulopathy, or localized or systemic infection

Ages: 19 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pain 3 months after surgery | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea